CLINICAL TRIAL: NCT05986240
Title: A Phase I Study Investigating the Safety & Efficacy of Danvatirsen as Monotherapy Followed by Combination With Venetoclax in Patients With Relapsed/Refractory MDS & AML
Brief Title: Danvatirsen Monotherapy Followed by Combination With Venetoclax in Relapsed/Refractory MDS & AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Flamingo Therapeutics NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14320; R01FD007836-01 (FDA)
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: AML/MDS; Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — danvatirsen; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Danvatirsen Monotherapy (Experimental): Patients will be enrolled in cohorts of 3 for the Danvatirsen dose escalation substudy. Based on the DLT of the first cohort of participants, subsequent cohorts will either be administered doses at the next higher dose level, de-escalated to the next lower dose level, or remain the same. Dose escalation discontinuations and MTD will be determined as described in the 'Detailed Study Description.' The total duration of 1 cycle is approximately 4 weeks (28 days). Proposed dose levels and treatment schedule are as follows:
  Dose Level 1 (DL1): Danvatirsen Day 1 - Day 28 (1mg/kg loading dose on Cycle 1/Day 1 (C1D1), Cycle 1/Day 3 (C1D3); and Cycle 1/Day 5 (C1D5) followed by weekly 1mg/kg infusion for 3 weeks) Dose Level 2 (DL2): Danvatirsen Day 1 - Day 28 (2mg/kg loading dose on C1D1, C1D3, and C1D5 followed by weekly 2mg/kg infusion for 3 weeks) Dose Level 3 (DL3): Danvatirsen Day 1 - Day 28 (3mg/kg loading dose on C1D1, C1D3, and C1D5 followed by weekly 3mg/kg infusion for 3 weeks)
  Interventions: Drug: Danvatirsen
- Danvatirsen + Venetoclax Combination Therapy (Experimental): Patients will be enrolled in cohorts of 3 for the Danvatirsen + Venetoclax dose escalation substudy. Dose escalation administration will be as described in the Danvatirsen monotherapy substudy arm and dose escalation discontinuations and MTD will be determined as described in the 'Detailed Study Description.'
  Up to 2 dose levels of Danvatirsen will be evaluated based on data from the Danvatirsen monotherapy arm. Dose 1 will be one level lower than the dose with expected target activity.
  Venetoclax: 400 mg (or equivalent) administered as fixed dose daily (except for specific dose modifications described in the protocol) orally for 28 days per cycle. To mitigate risk of tumor lysis syndrome, during Cycle 1 Venetoclax will be dose escalated daily to the goal dose of 400mg daily (100mg on Day 1, 200mg on Day 2 and 400mg on Day 3, and onwards, or adjusted dose ramp-up per Venetoclax label if on concomitant azoles).
  The three cycles are approximately 28 days each in duration.
  Interventions: Combination Product: Danvatirsen + Venetoclax

INTERVENTIONS:
Drug: Danvatirsen — Danvatirsen (AZD9150) is a selective, high-affinity, antisense oligonucleotide inhibitor of signal transducer and activator of transcription 3 (or STAT3).
  Other Names: AZD9150
  Arms: Danvatirsen Monotherapy
Combination Product: Danvatirsen + Venetoclax — Danvatirsen (AZD9150) is a selective, high-affinity, antisense oligonucleotide inhibitor of signal transducer and activator of transcription 3 (or STAT3).
  Venetoclax: Commercially available. Venetoclax is a potent, selective small molecule inhibitor of BCL-2, an anti-apoptotic protein found on some types of cancer cells.
  Other Names: Venclexta
  Arms: Danvatirsen + Venetoclax Combination Therapy

SUMMARY:
This is a Phase 1 study investigating the safety and efficacy of Danvatirsen as a monotherapy followed by combination with Venetoclax in patients with relapsed/refractory myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML).

Funding Source: FDA OOPD

DETAILED DESCRIPTION:
This is a Phase 1 study investigating the safety and efficacy of Danvatirsen as a monotherapy followed by combination with Venetoclax in patients with intermediate/high/very high myelodysplastic syndromes (MDS) as determined by revised International Prognostic Scoring System (IPSS-R) or acute myeloid leukemia (AML) who have relapsed or are refractory to frontline therapy. Danvatirsen is a next generation, high affinity, antisense oligonucleotide inhibitor of signal transducer and activator of transcription 3 (or STAT3) that has shown preclinical activity in vitro and good intracellular uptake in vivo in primary patient MDS and AML stem cells. STAT3 is a transcription factor that is overexpressed and dysregulated in several malignancies. Venetoclax is a commercially available, potent, selective small molecule inhibitor of B-cell Lymphoma-2 (BCL-2), an anti-apoptotic protein found on some types of cancer cells. Prior studies have demonstrated a strong correlation between STAT3 & Myeloid cell leukemia-1 (MCL-1) overexpression. MCL-1 is a multi-domain anti-apoptotic protein belonging to the BCL-2 family, which regulates the intrinsic apoptosis pathways and plays a central role in mediating therapeutic resistance to novel therapies such as Venetoclax in MDS and AML.

While FDA approved therapies have moved the field forward in newly diagnosed AML, relapsed/refractory (R/R) MDS and R/R AML continue to have a dismal prognosis, with a median overall survival of 4-10 months.

The study team has designed an innovative clinical trial to study Danvatirsen as monotherapy followed by combination with venetoclax for the treatment of relapsed/refractory high-risk MDS/AML. The study team plans to incorporate several important pharmacodynamic endpoints that will provide a real-time assessment of the effect of STAT3 inhibition in MDS/AML stem & progenitor cells and the impact on target gene expression. These correlative studies will help identify subsets of patients that are most likely to respond to STAT3 inhibition. Although direct targeting and monitoring of aberrant stem cells has recently gained some traction in AML, it is a novel approach for the treatment of MDS.

This study has been designed as a Phase 1 dose-escalation protocol of 2 different sub-studies to evaluate the safety profile, determine the Maximum Tolerated Dose (MTD) of Danvatirsen monotherapy followed by combination with Venetoclax once safety of Danvatirsen monotherapy is established. Patients with intermediate/high/very high IPSS-R MDS or AML who have relapsed/or are refractory to all available frontline therapy with no FDA approved treatment options will be enrolled in both the sub-studies. The objective of determining the MTD is to be able to find the minimum safe and biologically effective dose to be the recommended Phase 2 dose. For both the sub-studies safety, efficacy and assessment of PK/PD will be used to inform the recommended phase 2 dose.

Arms/Groups are detailed in the 'Arms/Groups' module of this record. Dose-escalation for each substudy is as follows:

Substudy 1 (Danvatirsen Monotherapy): The maximum number of patients to be enrolled in the dose-escalation phase for Danvatirsen monotherapy is 12, and patients will be treated in cohorts of 3. Based upon study parameters for Bayesian Optimal Interval (BOIN) design with a target Dose Limiting Toxicity (DLT) rate of 25%, if the observed DLT rate at the current dose ≤ 0.197, the next cohort of patients will be treated at the next higher dose. If it is > 0.298, dosing will be de-escalated to the next lower dose level. Otherwise, the next cohort of patients will be enrolled at the current dose. Dose escalation will discontinue and the Maximum Tolerated Dose (MTD) will be determined: (1) once all patients have been enrolled, (2) 6 patients have been treated at the same dose level with the decision to stay, or (3) all doses are found to be too toxic. Patients that were not evaluable for Dose Limiting Toxicities (DLTs) will be replaced. To accrue 12 evaluable patients, up to 20 patients will probably have to be entered, and this will take 2 years to complete. The total duration of 1 cycle is approximately 4 weeks (28 days).

Substudy 2 (Danvatirsen + Venetoclax Combination): The maximum number of patients to be enrolled in the dose-escalation phase for Danvatirsen + Venetoclax combination is 12, and patients will be treated in cohorts of 3. Based upon the study parameters for BOIN design with target DLT rate of 25%, if the observed DLT rate at the current dose ≤ 0.197, the next cohort of patients will be treated at the next higher dose. If it is > 0.298, dosing will be de-escalated to the next lower dose level. Otherwise, the next cohort of patients will be enrolled at the current dose. Dose escalation for the combination therapy will discontinue and Maximum Tolerated Dose (MTD) will be determined: (1) once all 12 patients have been enrolled, (2) 9 patients have been treated at the same dose level with the decision to stay, or (3) all doses are found to be too toxic. To accrue 12 evaluable patients, up to 18 patients will have to be enrolled, and this will take about one and half years to complete. The total duration of 1 cycle is again approximately 4 weeks (28 days).

Dose Modifications (referenced in 'Arms/Groups'):

Dose modification guidelines apply to both sub-studies and are minimal recommendations. Further reductions are permitted based on PI's clinical judgment following Sponsor approval.

In general, in the event of ≥ Grade 3 hematological toxicities, laboratory values should be monitored weekly (or more frequently until ≤ Grade 2).

Proposed dose modifications for treatment related toxicity (hematological) Worst Toxicity (CTCAE V5.0 Grade Recommended Dose Modification) Thrombocytopenia: Grade 4 (Platelet < 25,000/mm3) Dose delay until resolved to ≤ Grade 2

* If resolved to ≤ Grade 2 in ≤ 7 days, then maintain dose level
* If resolved to ≤ Grade 2 in > 7 but ≤ 21 days, then lower 1 dose level
* Permanently discontinue treatment if not resolved to ≤ Grade 3 in 21 days.

Proposed dose modifications for treatment related toxicity (non-hematological) Worst Toxicity (CTCAE V5.0 Grade Recommended Dose Modification) Grade 2: Dose delay until ≤ Grade 1 or baseline and maintain dose level Grade 3: Dose delay until resolved to ≤ Grade 1 or baseline

* If resolved in ≤ 7 days, then maintain dose level
* If resolved in > 7 days but ≤ 14 days, then lower 1 dose level
* If not resolved in ≤ 14 days, then permanently discontinue treatment Grade 4 : permanently discontinue treatment

Danvatirsen dose reductions Dose reduction for toxicity is allowed to one dose level below the current level. For the lowest dose of 1 mg/kg, dose reduction is allowed to 0.5 mg/kg below that dose level. Once a dose has been reduced for a given patient due to toxicity, this dose should be administered for all subsequent infusions, unless a further dose reduction is required. Any subsequent dose re-escalation would require consultation with the PI. Up to 1 dose level reduction is permitted.

Venetoclax Dose Modifications:

During cycle 1, Venetoclax will be dose escalated daily to the goal dose. Patients will receive 100mg on Day 1, 200mg on Day 2 and 400mg on Day 3 and onwards, or adjusted dose per venetoclax label if on concomitant azoles. The goal is to administer 28 days of venetoclax in cycle 1 unless marrow remission with concomitant marrow hypocellularity and/or myelosuppression is confirmed earlier than cycle 1 Day 28. In this case the venetoclax may be stopped earlier to avoid venetoclax related myelosuppression or further marrow hypo/aplasia after discussion and approval from the PI.

Initial response assessment will occur after 21 days of study therapy. Participants with stable or responding disease may continue on study until completion of study if their treating physician and PI feel that they are deriving clinical benefit. Participants with significant AEs or progressive disease or those having absence of clinical benefit after 6 cycles of treatment should be removed from study. Duration of therapy will depend on individual response, evidence of disease progression and tolerance. In the absence of significant adverse events, treatment may continue indefinitely or until one of the following criteria applies:

* Disease progression
* Intercurrent illness that prevents further administration of treatment
* Participant decides to withdraw from the study OR
* General or specific changes in the participant's condition or compliance render the participant unacceptable for further treatment in the opinion of the treating investigator.

All participants should undergo response evaluations between Day 21 and Day 42 of first and/or second induction course (optional). Unless there is clear evidence of progressive disease in the blood, bone marrow aspiration is required and bone marrow biopsy is strongly encouraged. In cases with hypocellular marrows (<10% cellularity), repeat bone marrow examinations should be considered when there is evidence of hematopoietic recovery. If multiple bone marrow examinations are performed, the last examination will be used to classify the patient's response. The final response will be determined no later than day 42 from the start of therapy. Clinical BMA should be repeated to assess response prior to cycles 3, 5 and 7 and subsequently after every 2 cycles of treatment and at the end of treatment for patients that initially responded

During treatment, all participants should undergo response evaluations prior to cycle 3. Unless there is clear evidence of progressive disease in the blood, bone marrow aspiration (BMA) is required and bone marrow biopsy is strongly encouraged. In cases with hypocellular marrows (<10 % cellularity), repeat bone marrow examinations should be considered when there is evidence of hematopoietic recovery. If multiple bone marrow examinations are performed, the last examination will be used to classify the patient's response. The final response will be determined no later than day 42 from the start of the first cycle of therapy. Clinical BMA should be repeated to assess response prior to cycles 3, 5 and 7 and subsequently after every 2 cycles of treatment and at the end of treatment for patients that initially responded.

When a participant discontinues the study, a final visit will be conducted. Following discontinuation of the study treatment, the participant will be treated according to the investigator's or treating physician's discretion. After the end-of-therapy visit, patients who have not progressed/relapsed or initiated subsequent anticancer therapy will be followed every 3 months for response assessment for up to 3 years, until the initiation of subsequent anticancer therapy, or until disease progression/relapse, whichever occurs first. All patients will be followed to document the start of subsequent anticancer therapy and overall survival (OS) every 3 months for up to 3 years after discontinuation of study drug. If a participant discontinues from the study due to an adverse event considered related to study treatment, a follow-up visit should be conducted no later than 30 days after the last dose of protocol therapy. Safety assessments are recommended at least every 14 days, until all toxicities resolve, return to baseline or become clinically satisfactory, stable, or are considered irreversible.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age at the time of signing the Informed Consent Form (ICF); must voluntarily sign an ICF; and be able to meet all study requirements
* Morphologically confirmed diagnosis of AML or MDS in accordance with World Health Organization (WHO) diagnostic criteria
* Subjects with relapsed/refractory AML who are refractory or relapsed to all conventional therapy and do not have any FDA approved or standard therapeutic options & subjects with intermediated/high/very high IPSS-R MDS who are refractory or relapsed to at least 2 cycles of hypomethylating agent based therapy (azacitidine / decitabine based) OR patients with rapid progression of disease regardless of number of cycles of therapy
* At least 3 months from Allogenic stem cell transplantation and no clinical sign of active graft vs host disease (GVHD)
* WBC must be <25,000 cells/uL and may be reduced with hydroxyurea to reach this goal prior to study start. Hydroxyurea can be administered on trial with an increase in WBC counts at the discretion of the PI
* A bone marrow biopsy must be performed within the screening window (day-28-day-1) and tissue collected for correlative analysis for entrance to this trial. Correlative sample collection is essential on this study
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Recovery to ≤ Grade 1 or baseline for any toxicities considered to be due to prior systemic treatments, excluding alopecia
* Must have adequate hepatic and renal function as follows:

ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN) or ≤ 5x ULN if considered to be leukemia related; Direct bilirubin ≤ 1.5 x ULN or ≤ 3x ULN (in patients with known Gilberts syndrome or if considered to be leukemia related)

* Serum creatinine clearance ≥ 45 mL/min/1.73 m2 either measured or calculated using standard Cockroft-Gault formula
* Subjects enrolled within childbearing ages of 18-50 years should use 2 forms of contraception while on study

Exclusion Criteria:

* Acute Promyelocytic Leukemia
* Low or very low risk MDS by IPSS-R after failure/progression of first line therapy with hypomethylating agents
* Active, uncontrolled infection. Patients with infection under active treatment and controlled with antibiotics are eligible. Use of prophylactic anti-microbials per institutional standards is allowed
* Active documented central nervous system (CNS) leukemia. Patients with a known history of CNS leukemia will be eligible if they have at least two most recent consecutive LPs showing clearance of CNS disease and no active/progressive symptoms thought to be related to the CNS disease
* Concurrent treatment with a non-permitted concomitant medication (as noted in protocol appendix)
* Concurrent anticancer treatment, major surgery, or the use of any investigational drug within 14 days before the start of trial treatment
* Other malignancy currently being treated or likely to need treatment in next 6 months with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ, surgically removed malignancies or malignancies definitively treated with chemotherapy, XRT and/or surgery with no evidence of active malignancy or not anticipated to need treatment in next 6 months or malignancies on maintenance therapy (e.g. tamoxifen for breast cancer) will be allowed after discussion and approval by both MPIs
* Pregnant or breastfeeding females
* Known current alcohol or drug abuse
* Clinically significant cardiovascular disease within the past 6 months (e.g. percutaneous intervention, coronary artery bypass graft, documented NYHA class III/IV cardiac heart failure, unstable angina or MI, poorly controlled atrial or ventricular arrhythmia) as determined by the investigator
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Legal incapacity or limited legal capacity to sign consent and/or participate in the trial
* Any condition deemed by the investigator to make the patient a poor candidate for clinical trial and/or treatment with investigational agents
* Previous exposure to the investigational agent (danvatirsen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Response to Therapy as determined by Overall Response Rate | From 21 days after initiation of study treatment to within 14 days following treatment discontinuation; up to 14 weeks total
  Overall Response Rate (ORR) will be used to assess clinical activity in AML and MDS participants. ORR will be measured as the percentage of participants demonstrating an objective overall response based upon a composite of remission related measures for AML and MDS participants as defined below.
  For AML participants, ORR will be defined as any confirmed Complete Remission (CR) + Complete Remission with Incomplete hematologic recovery (CRi) + Partial Remission (PR).
  or, AML = CR + CRi + PR
  For MDS participants, ORR will be defined as any confirmed Complete Remission (CR) + Complete Remission with Partial Hematologic Recovery (CRh) + Hematologic Response (HR).
  or, MDS = CR + CRh + HR
  Higher percentage is indicative of increased clinical activity of the danvatirsen monotherapy and danvatirsen + venetoclax combination therapies.

SECONDARY OUTCOMES:
Duration of Response | Up to 3 years after discontinuation of study treatment; up to 3.5 years total
  Duration of response will be measured by the number of days from the date of initial response (CRi or better) to the date of first documented disease progression/relapse or death, whichever occurs first. In the event that neither disease progression/relapse or death is documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, this endpoint will be censored at the date of last tumor assessment date. An increased duration of response is indicative of how long a patient will respond to treatment without tumor growth or metastasis
Event-free survival | Up to 3 years after discontinuation of study treatment; up to 3.5 years total
  Event-free survival (EFS) will be measured as the number of days from the date of treatment initiation to the date of documented treatment failure, relapse from complete remission, or death from any cause, whichever occurs first. In the event that none of the above are documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, this endpoint will be censored at the date of last tumor assessment date
Overall Survival | Up to 3 years after discontinuation of study treatment; up to 3.5 years total
  Overall Survival (OS) will be measured as the number of days from the date of treatment initiation until the date of death
30 Day All-cause mortality | 30 days after initiation of study treatment
  Number of participant deaths by all causes
60 Day All-cause Mortality | 60 days after initiation of study treatment
  Number of participant deaths by all causes

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Shastri, MBBS, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Montefiore Medical Center, The Bronx, New York
  - M.D. Anderson Cancer Center, Department of Leukemia, Houston, Texas

IPD SHARING:
Plan to Share IPD: No